CLINICAL TRIAL: NCT01185561
Title: A Pychoeducational Intervention for Women With Diabetes
Acronym: SWEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Sue Penckofer, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108324
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Anxiety; Anger
Keywords: Diabetes; SWEEP; Dysphoria
MeSH Terms: conditions — Depression; Anxiety Disorders; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual medical care (No Intervention): Participants assigned to this arm represent the control group and will receive usual medical care only.
- Psychoeducational intervention (Experimental): Participants assigned to this arm represent the experimental group and will receive group therapy for depression treatment based on cognitive behavioral therapy principles developed for women with type 2 diabetes
  Interventions: Behavioral: Psychoeducational intervention

INTERVENTIONS:
Behavioral: Psychoeducational intervention — The intervention is group therapy for depression treatment based on cognitive behavioral therapy principles developed for women with type 2 diabetes. Specifically, the intervention comprises activities including (1) Education about how dysphoric symptoms (i.e., depressive symptoms, anxiety, and anger) affect glycemic control; (2) Recognition of dysphoric symptoms; and (3) Management of dysphoric symptoms using cognitive-behavioral skills.
  Arms: Psychoeducational intervention

SUMMARY:
This proposal describes a small randomized study to determine whether usual medical care (UMC) for diabetes combined with a psychoeducational program is more effective than UMC for diabetes alone. This program differs from other diabetes programs by focusing on the management of dysphoric symptoms (depressive symptoms, anxiety, and anger). Diabetes self-care behaviors will be discussed and measured, but they are not the primary focus of the intervention. The psychoeducational program will address: 1) education about how dysphoric symptoms affect glycemic control; 2) recognition of dysphoric symptoms; and 3) management of dysphoric symptoms using Cognitive Behavioral Therapy (CBT). Subjects will be randomized to receive the group psychoeducational intervention or no additional treatment. All subjects will receive UMC for diabetes.

DETAILED DESCRIPTION:
Diabetes is the fifth deadliest disease in the United States with no known cure, and cardiovascular disease (CVD) is the leading cause of death in persons with diabetes. Diabetes is the only disease that causes women to have as much heart disease as men. The relative risk of cardiac mortality has been reported to be 2.6 for women with diabetes as compared to 1.9 for men with diabetes after controlling for other cardiac risk factors. While cardiac mortality for men with diabetes has declined (13.1%), there has been a 23% increase in age-adjusted cardiac mortality for women with diabetes. This poor outcome, occurring in a time of significant advances in the management of heart disease, suggests the need to consider directing treatment at other risk factors. Depression may be one such risk factor.

Depression is an independent risk factor for CVD, and is associated with poorer self-management and decreased health-related quality of life. Approximately 25% of persons with diabetes have depression, and the rate of depression in women with diabetes is double that of men with diabetes. Women with diabetes exhibit worse diabetes self-care, glycemic control, and poorer quality of life than men with diabetes, which are exacerbated by depression. Other affective symptoms including anxiety and anger commonly accompany depressive symptoms appear to impose similar risks for poor medical outcomes, and occur more often in women with diabetes than men with diabetes.

Research has shown that treatment of depression with medication and/or cognitive behavioral therapy (CBT) effectively relieves depression and improves glycemic control in persons with diabetes. More recent evidence suggests that these benefits are more durable in patients treated with CBT vs. antidepressants alone. There has been no research on "symptom clusters" (i.e., depression, anxiety, and anger) in persons with diabetes, and their effect on glycemic control and self-management. In addition, a CBT program to treat a cluster of dysphoric symptoms has not been tested in persons with diabetes. Since women with diabetes have greater depression and anxiety, worse glycemic control, and increased cardiac mortality than men with diabetes, we are proposing to test the feasibility and effectiveness of a psychoeducational intervention to promote emotional health in women with type 2 diabetes.

This proposal describes a small randomized controlled trial to determine whether usual medical care (UMC) for diabetes combined with a psychoeducational program is more effective than UMC for diabetes alone. This program differs from other diabetes programs by focusing on the management of dysphoric symptoms (depressive symptoms, anxiety, and anger). Diabetes self-care behaviors will be discussed and measured, but they are not the primary focus of the intervention. The psychoeducational program will address: 1) education about how dysphoric symptoms affect glycemic control; 2) recognition of dysphoric symptoms; and 3) management of dysphoric symptoms using CBT. A repeated measures, experimental design will be used. Subjects will be randomized to receive the group psychoeducational intervention or no additional treatment. All subjects will receive UMC for diabetes. The aims and hypotheses for the study are:

Primary Aim: To determine the effect of a psychoeducational intervention on dysphoric symptoms. The primary hypothesis is that women receiving a psychoeducational intervention plus UMC will report fewer dysphoric symptoms (depression, anxiety, and anger) at three and six months follow-up.

Secondary Aim: To determine the effect of a psychoeducational intervention on glycemic control, diabetes self-management, and health-related quality of life. The secondary hypothesis is that women receiving a psychoeducational intervention plus UMC will have decreased hemoglobin A1c, report better diabetes self-management (increased self-care behaviors and self-efficacy), and report increased health-related quality of life (increased functional status, life satisfaction, and decreased diabetes-related distress) at three and six months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 75 years;
2. have type 2 diabetes greater than six months and being medically managed
3. score greater than or equal to 16 on the Center for Epidemiological Studies Depression (CES-D) scale which is indicative of depressive symptoms.
4. score greater than or equal to 12 on the CES-D plus a history of depression or currently being treated for depression.

Exclusion Criteria:

Women with current alcohol or substance abuse disorders, or a history of bipolar depression or any other psychotic disorder will be excluded.

Women will also be excluded if they have a diabetes knowledge test score of less than 70% and severe complications of diabetes (blindness, renal failure, or major amputation which includes most toes, foot, knee, or leg)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Penckofer, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between March 2007 and November 2009
Pre-assignment Details: Eighty-four participants consented to participate in the study. Among these individuals, 10 (11.90%) were not randomized and were excluded from continuing their participation in the study because the medical monitor determined they had a significant psychiatric history, had a history of alcohol or drug abuse, or were not depressed.
Period: Overall Study
Arm/Group | Usual Medical Care | Psychoeducational Intervention
Started | 36 | 38
Completed | 34 | 26
Not Completed | 2 | 12
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 2 | 8

BASELINE CHARACTERISTICS:
Population: All randomized participants are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychoeducational Intervention | Usual Medical Care | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (8.8) | 54.0 (8.4) | 54.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 74
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: pounds (lbs)] | 229.1 (64.4) | 226.9 (48.7) | 228.0 (56.9)
Years Living with Diabetes [Mean (Standard Deviation); unit: years] | 10.5 (8.2) | 10.0 (6.5) | 10.3 (7.4)
CES-D [Mean (Standard Deviation); unit: units on a scale] — The CES-D is a self-report questionnaire assessing frequency and severity of depression symptoms. Scores may range from 0 to 60, where higher scores indicate worse mood.
  units on a scale | 27.7 (9.3) | 28.9 (9.5) | 28.3 (9.4)
STAI Trait Anxiety Subtest [Mean (Standard Deviation); unit: units on a scale] — The STAI trait anxiety subtest is a 20-item scale measuring state anxiety. Scores may range from 20 to 80 with higher scores indicating greater state anxiety.
  units on a scale | 51.6 (9.8) | 50.4 (9.2) | 51.0 (9.4)
STAI State Anxiety Subtest [Mean (Standard Deviation); unit: units on a scale] — The STAI state anxiety subtest is a 20-item scale measuring state anxiety. Scores may range from 20 to 80 with higher scores indicating greater state anxiety.
  units on a scale | 45.8 (12.8) | 47.9 (11.9) | 46.8 (12.3)
STAXI Anger Expression Subtest [Mean (Standard Deviation); unit: units on a scale] — The STAXI anger expression subtest is a 24-item scale measuring how anger is generally being experienced and expressed. Scores may range from 0 to 72 with higher scores indicating greater anger.
  units on a scale | 40.6 (13.2) | 34.7 (13.9) | 37.7 (13.8)

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies Depression (CES-D) Score
Description: The CES-D score was compared between those assigned to intervention versus those assigned to usual medical care six months after randomization. The CES-D is a self-report questionnaire assessing frequency and severity of depression symptoms. Scores may range from 0 to 60, where higher scores indicate worse mood.
Time Frame: 6 Months
Population: This analysis is restricted to participants who completed the final study visit six months after randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychoeducational Intervention | Usual Medical Care
Number analyzed (Participants) | 26 | 34
units on a scale | 12.6 (8.0) | 21.5 (10.2)
Statistical Analysis 1: Comparison: Psychoeducational Intervention vs Usual Medical Care; The null hypothesis is that there is no difference in CES-D score between those assigned to the psychoeducational intervention and those assigned to usual medical care six months after randomization; Test type: Superiority or Other; p = .001, t-test, 2 sided; Mean Difference (Final Values) = 8.89, 95% CI 2-sided [4.03 to 13.76], Standard Error of Mean 2.43

2. Secondary Outcome: State-Trait Anxiety Inventory (STAI Form Y-1) State Anxiety Sub-test Score
Description: Scores on the The State-Trait Anxiety Inventory (STAI Form Y-1) State Anxiety Sub-test are compared between those assigned to intervention versus those assigned to usual medical care six months after randomization. The STAI state anxiety subtest is a 20-item scale measuring state anxiety. Scores may range from 20 to 80 with higher scores indicating greater state anxiety.
Time Frame: 6 Months
Population: This analysis is restricted to participants who completed the final study visit six months after randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychoeducational Intervention | Usual Medical Care
Number analyzed (Participants) | 26 | 34
units on a scale | 35.7 (12.4) | 43.6 (12.6)
Statistical Analysis 1: Comparison: Psychoeducational Intervention vs Usual Medical Care; The null hypothesis is that there is no difference in the State Anxiety Sub-test score between those assigned to the psychoeducational intervention and those assigned to usual medical care six months after randomization; Test type: Superiority or Other; p = .02, t-test, 2 sided; Mean Difference (Final Values) = 7.82, 95% CI 2-sided [1.29 to 14.37], Standard Error of Mean 3.27

3. Secondary Outcome: State-Trait Anxiety Inventory (STAI Form Y-1) Trait Anxiety Sub-test Score
Description: Scores on the The State-Trait Anxiety Inventory (STAI Form Y-1) Trait Anxiety Sub-test are compared between those assigned to intervention versus those assigned to usual medical care six months after randomization. The STAI trait anxiety subtest is a 20-item scale measuring state anxiety. Scores may range from 20 to 80 with higher scores indicating greater state anxiety.
Time Frame: 6 Months
Population: This analysis is restricted to participants who completed the final study visit six months after randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychoeducational Intervention | Usual Medical Care
Number analyzed (Participants) | 26 | 34
units on a scale | 36.9 (10.1) | 45.3 (12.0)
Statistical Analysis 1: Comparison: Psychoeducational Intervention vs Usual Medical Care; The null hypothesis is that there is no difference in the State Trait Anxiety Sub-test score between those assigned to the psychoeducational intervention and those assigned to usual medical care six months after randomization; Test type: Superiority or Other; p = .005, t-test, 2 sided; Mean Difference (Final Values) = 8.48, 95% CI 2-sided [2.64 to 14.31], Standard Error of Mean 2.91

4. Secondary Outcome: State-Trait Anger Expression Inventory (STAXI) Anger Expression Sub-test Score
Description: Scores on the The State-Trait Anger Expression Inventory (STAXI) Anger Expression Sub-test will be compared between those assigned to intervention versus those assigned to usual medical care six months after randomization. The STAXI anger expression subtest is a 24-item scale measuring how anger is generally being experienced and expressed. Scores may range from 0 to 72 with higher scores indicating greater anger.
Time Frame: 6 Months
Population: This analysis is restricted to participants who completed the final study visit six months after randomization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychoeducational Intervention | Usual Medical Care
Number analyzed (Participants) | 26 | 34
units on a scale | 28.9 (13.7) | 29.6 (14.9)
Statistical Analysis 1: Comparison: Psychoeducational Intervention vs Usual Medical Care; The null hypothesis is that there is no difference in the State Trait Anger Expression Sub-test score between those assigned to the psychoeducational intervention and those assigned to usual medical care six months after randomization; Test type: Superiority or Other; p = .85, t-test, 2 sided; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-6.77 to 8.24], Standard Error of Mean 3.75

ADVERSE EVENTS:
Time Frame: Adverse data were collected for 2 years, 8 months
Arm/Group | Psychoeducational Intervention | Usual Medical Care
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/36
Other Adverse Events (participants affected / at risk) | 2/38 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychoeducational Intervention (N=38) | Usual Medical Care (N=36)
Inpatient Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — One patient was admitted inpatient for an acute stress reaction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychoeducational Intervention (N=38) | Usual Medical Care (N=36)
Worsening mood (Psychiatric disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes